CLINICAL TRIAL: NCT00079092
Title: A Phase II Trial Of Thalidomide And Procarbazine In Adults With Recurrent/Progressive Gliomas
Brief Title: Thalidomide and Procarbazine in Treating Patients With Recurrent or Progressive Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: REBACDR0000354204; CCCWFU-91202; NCI-6358
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult glioblastoma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Astrocytoma; Oligodendroglioma; Glioblastoma; Glioma; Gliosarcoma | interventions — Procarbazine; Thalidomide

INTERVENTIONS:
Drug: procarbazine hydrochloride
Drug: thalidomide

SUMMARY:
RATIONALE: Thalidomide may stop the growth of malignant glioma by stopping blood flow to the tumor. Drugs used in chemotherapy, such as procarbazine, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining thalidomide with procarbazine may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving thalidomide together with procarbazine works in treating patients with recurrent or progressive malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with recurrent or progressive malignant glioma treated with thalidomide and procarbazine.

Secondary

* Determine the progression-free survival of patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral procarbazine once daily on days 1-5 and oral thalidomide once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and then before every odd course.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 23-55 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioma

  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Glioblastoma multiforme
  * Anaplastic mixed oligoastrocytoma
* Progressive or recurrent disease* after radiotherapy with or without chemotherapy NOTE: *Patients with prior low-grade glioma who progressed after therapy and are found to have high-grade glioma are eligible
* Measurable disease by MRI or CT scan

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* More than 2 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* Transaminases ≤ 4 times upper limit of normal

Renal

* Creatinine ≤ 1.7 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 1 highly active method and 1 additional effective method of contraception for 1 month before, during, and for 4 weeks after study treatment
* No concurrent serious infection
* No other concurrent medical illness that would preclude study treatment
* No other malignancy within the past 5 years except curatively treated carcinoma in situ of the cervix or basal cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior thalidomide
* No concurrent prophylactic filgrastim (G-CSF)

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No prior procarbazine
* No more than 2 prior chemotherapy regimens for malignant glioma

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 3 months since prior radiotherapy

Other

* Recovered from prior therapy
* More than 7 days since prior antidepressants (selective serotonin reuptake inhibitors and/or monamine oxidase inhibitors)
* No concurrent antidepressants
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2004-01-01 (Actual); Primary Completion 2006-03-21 (Actual); Study Completion 2006-03-21 (Actual)

PRIMARY OUTCOMES:
Response rate by CT scan and MRI at baseline, pre-odd cycles, and study completion

SECONDARY OUTCOMES:
Progression-free survival by CT scan, MRI, and follow up form at baseline, pre-odd cycles, and study completion
Overall survival by follow-up form at study completion
Quality of life by FACT-Br, FACIT-F and Karnofsky performance status (PS) at baseline, pre-odd cycles, and study completion
Toxicity by evaluation form at baseline, pre-odd cycles, and study completion

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J. Lesser, MD, Principal Investigator — Wake Forest University Health Sciences; Edward G. Shaw, MD, Study Chair — Wake Forest University Health Sciences; Volker W. Stieber, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (5):
- United States (5):
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina